CLINICAL TRIAL: NCT05304858
Title: Connecting Lineage Target Expression and Immune Tumor Microenvironment Analysis of Prostate Cancer Metastasis
Brief Title: Tumor Microenvironment Analysis of Prostate Cancer Metastasis
Status: Recruiting | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: Janssen Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Mark Stein, Associate Professor of Medicine at the Columbia University Medical Center, Columbia University
Other Study IDs: AAAT2169
Record Dates: First submitted 2022-03-22; First posted 2022-03-31 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Recurrent Prostate Cancer
Keywords: Metastasis; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis | interventions — Biopsy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — In this study, researchers may perform whole genome sequencing and RNA sequencing on tissue samples.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TME Analysis: Participants who have been diagnosed with metastatic castration-resistant prostate cancer (mCRPC) will volunteer for a biopsy of a site in the body that contains prostate cancer, such as a bone, a lymph node or an organ such as the liver OR are planned to undergo standard of care surgical procedures such as orthopedic surgery or neurosurgery based on a subjects clinical needs.
  Interventions: Procedure: Biopsy

INTERVENTIONS:
Procedure: Biopsy — Standard of care surgical procedures to collect prostate cancer tissue from men with metastatic prostate cancers. Non-experimental.

SUMMARY:
The purpose of this study is to collect prostate cancer tissue from males with metastatic prostate cancers in order to study the tumor microenvironment (TME), which is the area surrounding the tumor including cells, blood vessels, etc., in men with metastatic prostate cancer. The type of research performed on these tissue samples include genetic & molecular analyses.

DETAILED DESCRIPTION:
The overall aim of this protocol is to collect prostate cancer tissue from males with metastatic prostate cancers in order to perform comprehensive profiling of the tumor microenvironment (TME) across sites of metastasis in males with metastatic prostate cancer. The TME is comprised of proliferating tumor cells, the tumor stroma, blood vessels, infiltrating inflammatory cells and a variety of associated tissue cells. This study will enable analysis of the prostate TME in the context of different sites of metastasis as well as a variety of clinical states of disease (i.e no prior androgen deprivation therapy, progression on abiraterone, progression on an androgen receptor (AR) antagonist, or progression on chemotherapy etc). Furthermore, the expression and receptor density of prostate lineage antigens that can be targeted for development of novel therapeutics for prostate cancer will be evaluated in parallel.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent for the trial.
* Age ≥18 years of age on day of signing informed consent.
* Eastern Cooperative Oncology Group (ECOG) performance status: 0,1 or 2
* Histologically proven adenocarcinoma of the prostate. (Rarely pathology is not available but if clinical situation confirms prostate cancer - such as prior response to androgen ablation and/or metastatic disease typical of prostate cancer, i.e. involving bone or pelvic/extra pelvic lymph nodes or para-aortic lymph nodes, AND an elevated serum concentration of prostate-specific antigen (PSA) typical of prostate cancer) pathology is not required and patient can be enrolled after discussed with study PI.
* Clinical stage N1 or M1
* Evidence of nodal or distant metastasis by MRI/CT scan, bone scan or positron emission tomography (PET) scan
* Planned specimen from subjects that undergo core needle biopsy must allow for cores of at least 21 gauge with depth of 5 mm. A goal of 3-8 core specimens (3 to 8 passages of the needle into the lesion) will be sought during the procedure, if felt to be safe by the performing physician.
* Laboratory tests meet minimum safety requirements:
* Hemoglobin >7mg/dL
* Platelet count ≥75,000/mm3
* Coagulation: prothrombin time (PT)/international normalized ratio (INR), Partial thromboplastin time (PTT) ≤ 1.5 upper limit of normal (ULN) (except if on therapeutic anticoagulation in which case the patient can be enrolled if stable and anticoagulation levels are appropriate for their condition per good clinical practice).

Exclusion Criteria:

* A psychiatric disorder, medical condition, or other life circumstance, which in the opinion of the investigators, would make it difficult for a patient to successfully complete the informed consent process.
* Acute illness or any medical condition in the judgment of the study physician making specimen collection inadvisable

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male adults age 18 or older diagnosed with metastatic castration-resistant prostate cancer (mCRPC).
Sampling Method: Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2021-09-15 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Single-Cell RNA Sequencing (scRNAseq) | 2 years
  Profiling of the tumor microenvironment (TME) through single-cell RNA sequencing (scRNAseq) for deep profiling of the local immune microenvironment in the tumor.
CyTOF high-parametric mass cytometry | 2 years
  CyTOF high-parametric mass cytometry for comprehensive profiling of the tumor and the tumor-immune microenvironment at a larger scale.
Multiplex Immunofluorescence | 2 years
  Multiplex immunofluorescence using Vectra multispectral microscope for high throughput spatial analysis of the tumor microenvironment.
Characterization of the expression and receptor density of prostate lineage antigens | 2 years
  Tumor tissue will be examined through genetic tests in order to determine gene expression of the tumor cells

CONTACTS AND LOCATIONS:
Overall Officials: Mark N. Stein, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No